CLINICAL TRIAL: NCT05109884
Title: Comparison of PET Imaging Patterns With Prostate-specific Membrane Antigen and Androgen Specific Receptor Expression Patterns in Prostate Cancer and Bladder Cancer
Brief Title: Comparison of PET Imaging Patterns With PSMA and AR Expression in Prostate Cancer and Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Markus Zeitlinger, Principal Investigator, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PC_LBI:AD_V3
Record Dates: First submitted 2021-09-28; First posted 2021-11-05 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- newly diagnosed very high risk locally advanced and/or oligometastatic prostate cancer (Other)
  Interventions: Diagnostic Test: PSMA PET Scan; Diagnostic Test: FDHT PET Scan
- metastatic, castration resistant prostate cancer (Other)
  Interventions: Diagnostic Test: PSMA PET Scan; Diagnostic Test: FDHT PET Scan
- newly diagnosed prostate cancer with planned radical prostatectomy (Other)
  Interventions: Diagnostic Test: PSMA PET Scan; Diagnostic Test: FDHT PET Scan
- primary bladder cancer with planned radical cystectomy (Other)
  Interventions: Diagnostic Test: PSMA PET Scan; Diagnostic Test: FDHT PET Scan

INTERVENTIONS:
Diagnostic Test: PSMA PET Scan — [68Ga]Ga-PSMAHBED-CC (Ga-PSMA) PET Scan
Diagnostic Test: FDHT PET Scan — [18F]-fluoro-5α-dihydrotestosterone (18F-FDHT) PET Scan

SUMMARY:
Patients suffering either from newly diagnosed very high risk locally advanced and/or oligometastatic prostate cancer (cohort A), metastatic castration-resistant prostate cancer (mCRPC, cohort B), newly diagnosed postate cancer with planned radical prostatectomy (cohort C) or primary bladder cancer with planned radical cystectomy (cohort D) as identified by a multidisciplinary team of specialists, will be included.

PET imaging patterns using PSMA- and FDHT PET scans will be correlated with prostate-specific membrane antigen and androgen specific receptor expression patterns in prostate cancer and bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* Age 18-75 years
* Histologically or cytologically confirmed adenocarcinoma of the prostate with very high risk for the development of metastases (defined as PSA ≥20 or Gleason Score ≥8 or ≥cT3) and/or oligometastatic (T any, N positive, M any or T any, N any, M positive)
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade 0 or 1
* Planned radical prostatectomy
* ≤ 5 osseous metastasis
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, and other study procedures

Cohort B - mCRPC:

* Age ≥ 18 years
* Histologically or cytologically confirmed prostate adenocarcinoma.
* Presence of skeletal or nodal metastases according to one of the following criteria:
* Confirmed pathological fracture related to the disease OR
* Confirmation of distant bone and/or nodal metastases on CT or MRI scan or bone scintigraphy.

OR

* Positive pathology report of metastatic lesion.
* Disease progression despite ADT as indicated by:
* PSA increase that is ≥ 2 ng/mL and ≥ 25% above the minimum PSA as reached during ADT or above the pre-treatment level, if no response was observed and which is confirmed by a second value 1 or more weeks later.

OR

* Progression of measurable lymph nodes (short axis ≥ 15 mm) or visceral lesion measurable per RECIST OR
* New metastatic lesions appearing on bone scan/imaging
* Chemical or surgical castration
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, and other study procedures

Cohort C:

* Age ≥ 18 years
* Histologically or cytologically confirmed prostate adenocarcinoma.
* Planned radical prostatectomy
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, and other study procedures

Cohort D:

* Age ≥ 18 years
* Histologically or cytologically confirmed bladder cancer.
* Planned radical cystectomy
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study participation
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory and radiographic assessments, and other study procedures

Exclusion Criteria:

Cohort A:

* Tumour infiltration of the rectum or pelvic wall
* Visceral metastasis
* HIV positive
* Any contraindication for surgery
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan (if applicable)
* Patient's not eligible for the size of the PET/MRI gantry

Cohort B - mCRPC:

* HIV positive
* Any contraindication for tissue biopsy (if tissue biopsy is planned)
* Any contraindication for surgery (if surgery is planned)
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan (if applicable)
* Patient's not eligible for the size of the PET/MRI gantry

Cohort C:

* Any contraindication for surgery
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan (if applicable)
* Patient's not eligible for the size of the PET/MRI gantry

Cohort D:

* Any contraindication for surgery
* Any other condition that, in the opinion of the Investigator, would impair the patient's ability to comply with study procedures.
* Any contraindication for performing a PET/MRI scan (if applicable)
* Patient's not eligible for the size of the PET/MRI gantry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Correlation of PET imaging parameters with PSMA and AR expression levels | through study completion, an average of 3 years
  To correlate PET imaging parameters with prostate-specific membrane antigen (PSMA), and androgen specific receptor expression levels in tissue biopsy samples using immuno-histochemical methods (IHC).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No